CLINICAL TRIAL: NCT06603220
Title: An Open Label Study Evaluating the Safety, Tolerability, and Efficacy of EVO756 in Adults With Chronic Inducible Urticaria
Brief Title: A Study Evaluating the Safety, Tolerability, and Efficacy of EVO756 in Adults With Chronic Inducible Urticaria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Evommune, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EVO756-CIU001
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Chronic Inducible Urticaria
Keywords: chronic inducible urticaria; inducible urticaria
MeSH Terms: conditions — Chronic Inducible Urticaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- EVO756 (Experimental)
  Interventions: Drug: Oral EVO756

INTERVENTIONS:
Drug: Oral EVO756 — Oral EVO756, once daily

SUMMARY:
This phase 2a trial will evaluate the safety and efficacy of EVO756 in subjects with chronic inducible urticaria, including symptomatic dermographism and cold urticaria.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of chronic inducible urticaria for at least 3 months.
* Positive response following provocation using the TempTest or FricTest at Screening and Day 1.

Exclusion Criteria:

* History of diseases other than chronic inducible urticaria or chronic spontaneous urticaria with urticaria or angioedema symptoms, such as urticarial vasculitis, erythema multiforme, cutaneous mastocytosis (urticaria pigmentosa), and hereditary or acquired angioedema.
* Concurrent use of certain medications, including antihistamines.
* Any clinically significant disease, or other skin disease or skin markings (e.g., extensive scarring, tattoos), that might confound the evaluation of safety or efficacy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-08-14 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | Day 1 to Week 6
  Safety will be assessed through an evaluation of treatment emergent adverse events, physical exams, vital signs, laboratory tests, and 12-lead ECGs.

SECONDARY OUTCOMES:
Change in Total Fric Score (TFS) | Day 1 to Week 4
  Changes in the number of prongs that elicit a wheal response using a FricTest for subjects with symptomatic dermographism.
Change in Critical Temperature Threshold (CTT) | Day 1 to Week 4
  Changes in the highest temperature that elicits a wheal response using a TempTest for subjects with cold urticaria.
Change in pruritus severity at the provocation test site | Day 1 to Week 4
  Changes in the severity of pruritus at the provocation test site using an 11-point numerical rating scale.

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Cahaba Dermatology & Skin Health Center, LLC, Birmingham, Alabama
  - California Allergy and Asthma Medical Group, Los Angeles, California
  - Integrative Skin Science and Research, Sacramento, California
  - West Dermatology Research Center, San Diego, California
  - Advanced Clinical Research Institute, Tampa, Florida
  - Aeroallergy Research Laboratories of Savannah, Inc., Savannah, Georgia
  - Treasure Valley Medical Research, Boise, Idaho
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Southern Indiana Clinical Trials, New Albany, Indiana
  - Indiana Clinical Trials Center, P.C., Plainfield, Indiana
  - DelRicht Research, Baton Rouge, Louisiana
  - Chesapeake Clinical Research, Inc, White Marsh, Maryland
  - OptiSkin Medical, New York, New York
  - Red River Research Partners, Fargo, North Dakota
  - Bexley Dermatology Research, Bexley, Ohio
  - Allergy, Asthma, and Clinical Research Center, Oklahoma City, Oklahoma
  - Allergy and Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - Austin Institute for Clinical Research, Pflugerville, Texas